CLINICAL TRIAL: NCT06908369
Title: Persistent Cardiac Symptoms in Patients With Adequately Treated Graves' Disease
Brief Title: Cardiac Symptoms in Patients With Treated Graves' Disease
Acronym: CARD-GRAVES
Status: Active, not recruiting | Type: Observational
Sponsor: Ulla Feldt-Rasmussen (Other)
Responsible Party: Sponsor-Investigator, Ulla Feldt-Rasmussen, MD, DMSc, Professor Emerita, Senior Research Consultant, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: Cardiac Symptoms in Graves; Rigshospitalet, Capital Region (Other: Rigshospitalet, Capital Region of Denmark)
Record Dates: First submitted 2025-03-18; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Graves Disease; Cardiac Arrhythmias; Cardiac Structure and Function
MeSH Terms: conditions — Graves Disease; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 60 ml of blood is drawn and transferred to different test tubes with different chemical additives. The blood samples are used for determination of biochemical, hematological and immunochemical parameters in accordance with Rigshospitalet's LabPortal.
  3 x 9 ml of blood is drawn for genetic analyses. The blood is transferred to a glass with Ethylenediaminetetraacetic acid (EDTA) and glass with Trasylol and frozen and stored at -80 degrees.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with treated Graves' disease and cardiac symptoms: Patients with Graves' disease, who have been treated to biochemical euthyroidism but still experience cardiac symptoms.

SUMMARY:
Hyperthyroidism is a condition with increased production of thyroid hormone from the thyroid gland. Hyperthyroidism affects the heart's inotropy (contractile force) and chronotropy (rhythm). Therefore, patients often experience symptoms such as increased/irregular heart rate, pounding heartbeats, and shortness of breath. The cardiac symptoms often improve when hyperthyroidism is treated and biochemical euthyroidism is achieved. However, knowledge of the long-term effects on the heart is limited. Existing studies have generally shown that patients with hyperthyroidism have an increased morbidity and mortality.

The investigators conducted a questionnaire survey which showed that about 38% of patients with Graves' disease continue to experience cardiac symptoms even months after normalization of thyroid hormone concentrations in the blood. This observation supports the presence of a persistent cardiovascular dysfunction, which may be due to a modulation of genomic or non-genomic factors with an effect on the cardiovascular system. These reflections are the focus of this clinical study. The aim of the study is to investigate the possible pathophysiology for this new "syndrome" in biochemically euthyroid patients. It is not a repetition of previous similar experiments.

DETAILED DESCRIPTION:
Cardiac symptoms are common i patients with Graves' disease. These symptoms often disappear when hyperthyroidism is treated. However, a subgroup of patients with Graves' disease experiences persisting cardiac symptoms after treatment. The aim of the study is to describe these symptoms and investigate their origin.

A total of 75 patients are included in the study. Patients were recruited from the Department of Nephrology and Endocrinology at Copenhagen University Hospital Rigshospitalet and the Department of Internal Medicine, Section of Endocrinology at Herlev Gentofte Hospital, Denmark. The patients were identified by extracting a list of patients with the International Classification of Diseases 10 codes (ICD 10 codes) E050 and E059. Also, a list of patients with positive thyrotropin receptor antibody (TRAbI measurements was extracted.

All patients had a thorough cardiac work up including blood samples, 12-lead resting electrocardiogram, 24-hour electrocardiogram monitoring (Holter), transthoracic echocardiography, and exercise stress test. The focus was to investigate whether the cardiac symptoms could be explained by structural or functional changes of the heart or by cardiac arrhythmias.

All patients were questioned about their symptoms including: type of cardiac symptoms, frequency and when they occured. The focus was to gain knowledge on the clinical presentation of cardiac symptoms in the subgroup.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Graves' disease
* Between the ages of 18 and 55 years
* Has been euthyroid for at least three months prior to inclusion
* Experiences cardiac symptoms

Exclusion Criteria:

* Cardiovascular disease
* Deemed unsuitable by project staff (e.g. due to language problems)
* Pregnancy
* Alcohol abuse or other abuses

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants are recruited from the Endocrinology Outpatient Clinic at Rigshospitalet and Herlev/Gentofte Hospital.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Cardiac changes | The cardiac examinations were performed during three study visits which extended over a period of approximately half a year.
  The patients were examined for cardiac arrhythmias and structural and functional changes of the heart with resting 12-lead ECG, 24-hour ambulatory ECG monitoring, transthoracic echocardiography, and exercise stress test.
  ECG analyses included: heart rate, PR-interval, QRS-duration, and QT-interval. Any presence of abnormal cardiac axis, bundle branch block, atrioventricular (AV) block, ventricular hypertrophy or atrial enlargement was noted.
  Analysis of the 24-hour ECG recording including heart rate, detection of arrythmia, heart block, and reported symptoms.
  The echocardiographic analysis consisted of the following measurements: left ventricular dimensions, left ventricular volumes, left ventricular function, left atrial volume, right ventricular dimensions, right ventricular function, and pulmonary artery pressure.
  Analysis of the exercise stress test included blood pressure, heart rate, and ECG-changes indicating myocardial ischemia and arrhythmias.

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Feldt-Rasmussen, MD; DMSc, Study Director — Rigshospitalet, Denmark; Stig Haunsø, MD; DMSc, Study Director — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

DOCUMENTS (1):
  • Study Protocol (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT06908369/Prot_000.pdf